CLINICAL TRIAL: NCT06888479
Title: Optimal Timing of Hepatitis B Vaccination After Transplants: a Randomized Clinical Study
Brief Title: Optimal Timing of Hepatitis B Vaccination After Transplants
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IIT2024061
Record Dates: First submitted 2025-01-14; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Transplant-Related Disorder; Hepatitis B Virus Infection; Vaccine Reaction
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 'Early Vaccination' (low-risk) (Experimental): Patients with composite immune risk score (CIRS) ≤ 2.5 and being assigned to receive 3 doses of hepatitis B vaccine at 3, 4, and 9 months after transplantation.
  Interventions: Biological: hepatitis B vaccine
- 'Early Vaccination' (high-risk) (Experimental): Patients with CIRS > 2.5 and being assigned to receive 3 doses of hepatitis B vaccine at 3, 4, and 9 months after transplantation.
  Interventions: Biological: hepatitis B vaccine
- 'Guideline' (low-risk) (Active Comparator): Patients with CIRS ≤ 2.5 and being assigned to receive 3 doses of hepatitis B vaccine at 6, 7, and 12 months after transplantation.
  Interventions: Biological: hepatitis B vaccine
- 'Guideline' (high-risk) (Active Comparator): Patients with CIRS > 2.5 and being assigned to receive 3 doses of hepatitis B vaccine at 6, 7, and 12 months after transplantation.
  Interventions: Biological: hepatitis B vaccine

INTERVENTIONS:
Biological: hepatitis B vaccine — Three doses of hepatitis B vaccine

SUMMARY:
The investigators aim to perform a randomized clinical trial to determine the optimal timing of hepatitis B vaccination after hematopoietic cell transplantation (HCT) through evaluating the immunity effect of two different vaccination schedules (initiated at 3 or 6 months after transplantation) in patients with different immune reconstitution status.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥ 16 years old;
2. Patients receiving hematopoietic cell transplantation;
3. Patients achieving complete molecular remission;
4. Patients or their guardians have to sign an informed consent form before the start of the research procedure.

Exclusion Criteria:

1. Multiple transplantations;
2. Donors' HBV-DNA or HBsAg are positive;
3. Patients' HBV-DNA or HBsAg are positive before transplantation or < 3 months after transplantation;
4. Patients who are unable to comply with the research treatments and monitoring requirements due to mental or other medical conditions;
5. Patients who are ineligible for the study due to other reasons which would cause unacceptable risks to the patients.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Titer of hepatitis B surface antibodies (HBsAb). | One month after the completion of 3 doses of hepatitis B vaccine.
  The investigators will compare the titer of HBsAb one month after the completion of 3 doses of hepatitis B vaccine in transplants with different timing of hepatitis B vaccination, different donor type and different immune reconstitution status.

SECONDARY OUTCOMES:
HBV infection | Through study completion, an average of 1 year
  HBV-DNA or HBsAg are positive

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes